CLINICAL TRIAL: NCT06760793
Title: Comparison of the Effectiveness of Static Stretching and Deep Friction Massage Applied to Plantar Flexors in Children With Spastic Cerebral Palsy
Brief Title: Deep Friction Massage in Children With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Meltem Koc, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/30
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Spastic Cerebral Palsy (sCP)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental)
  Interventions: Other: manual static stretching exercises on plantar flexors
- Group 2 (Experimental)
  Interventions: Other: deep friction massage on plantar flexors

INTERVENTIONS:
Other: manual static stretching exercises on plantar flexors — A manual static stretching exercises was performed on the plantar flexors in both knee extension and flexion. The stretch was applied while the participant was in a prone position
  Arms: Group 1
Other: deep friction massage on plantar flexors — Deep Friction Massage was applied to both the gastrocnemius muscle and the Achilles tendon. Participants were positioned in a prone posture for both applications
  Arms: Group 2

SUMMARY:
The aim of this clinical trial is to determine whether deep friction massage and stretching reduce muscle contraction in the calf muscle. The primary questions it seeks to answer are:

* Does deep friction massage or stretching reduce muscle contraction?
* Does deep friction massage or stretching improve walking?
* Does deep friction massage or stretching increase ankle joint range of motion?

Participants:

Participants will undergo either deep friction massage or stretching exercises for 10 minutes, three days a week, over a period of six weeks.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of spastic diplegic or hemiparetic CP
* aged between 3 and 18 years
* classified as level I, II, or III according to the Gross Motor Function Classification System (GMFCS)
* possessing sufficient cognitive function to cooperate.

Exclusion Criteria:

* Botulinum toxin (BoNT) injections to the lower extremity muscles within the last six months
* undergoing any surgery such as muscle lengthening or joint contracture within the last six months
* non-participation in two consecutive exercise sessions
* experiencing illnesses such as infections or musculoskeletal injuries during the study period.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
The Modified Ashworth Scale | before intervention and after 6 weeks
  The Modified Ashworth Scale (MAS) is the most widely used clinical scale for measuring increases in muscle tone. The original Ashworth Scale was a 5-point numerical scale that graded spasticity from 0 to 4, with 0 indicating no resistance and 4 indicating a limb that is rigid in flexion or extension.

SECONDARY OUTCOMES:
The Modified Tardieu Scale | Before intervention and after 6 weeks
  The Modified Tardieu Scale (MTS) is a clinical tool used to assess spasticity by evaluating the muscle's response to passive stretch at varying velocities. This scale was a 5-point numerical scale that graded spasticity from 0 to 5, with 0 indicating no resistance and 5 indicating a limb that is rigid in flexion or extension.
Range of motion (ROM) | Before intervention and after 6 weeks
  Range of motion (ROM) of ankle assessments were conducted using a standard goniometer. In these measurements, the initial position of the ankle was set to a 90° angle between the fibula and the 5th metatarsal. Participants were positioned in a supine position with a thin pillow placed under their knees. The pivot point of the goniometer was aligned with the lateral malleolus, while the fixed arm was positioned parallel to the midline of the fibula. The moving arm of the goniometer followed the midline of the 5th metatarsal. The participant was then instructed to perform active dorsiflexion and plantar flexion movements, with the results recorded. This procedure was repeated for passive dorsiflexion and plantar flexion movements
The Modified Timed Up and Go Test (TUG) | Before intervention and after 6 weeks
  The Modified Timed Up and Go Test (TUG) is a simple and objective clinical test that assesses walking speed, postural control, functional level, balance, and locomotor performance. In this test, the participant is asked to rise from a chair without armrests, walk at their own pace to touch a target placed 3 meters away, return to the starting point, and sit down again. The time taken to complete this task is recorded in seconds. The participant's starting position is sitting in a chair with the hip and knee joints flexed at 90°

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sitki Kocman University, Muğla, Menteşe, Turkey (Türkiye)